CLINICAL TRIAL: NCT07190170
Title: Time Restricted Eating for WeIght LoSs MainTenance-2 (TWIST-2): A Single-site, 2-arm Randomized Clinical Trial in Adults With Recent Weight Loss
Brief Title: Time Restricted Eating for WeIght LoSs MainTenance-2
Acronym: TWIST-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-00320; 4R00HL163474 (NIH)
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Weight Loss; Weight Gain; Weight Loss Maintenance
Keywords: obesity; time-restricted eating; weight-loss maintenance
MeSH Terms: conditions — Weight Loss; Weight Gain; Obesity; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-Restricted Eating (TRE) (Experimental): Participants assigned to the intervention: ≤10-hour/day time restricted eating.
  Interventions: Behavioral: TRE
- Baseline Advice Control (CON) (Active Comparator): Participants assigned to receive baseline advice.
  Interventions: Behavioral: Weight-Loss Maintenance Advice

INTERVENTIONS:
Behavioral: TRE — Participants randomized to the TRE arm will be instructed to consume all food and beverages in a self-selected 10-hr eating window.
  Arms: Time-Restricted Eating (TRE)
Behavioral: Weight-Loss Maintenance Advice — The CON arm participants will receive written baseline advice following randomization assignment that includes determinants associated with long-term weight-loss maintenance success (e.g., physical activity, and strategies to limit calorie intake).
  Arms: Baseline Advice Control (CON)

SUMMARY:
The TWIST 2.0 Study is a 12-month, 2-arm RCT in adults with recent weight loss. We will examine the efficacy of TRE on weight (Aim 1a) and fat mass (Aim 1b) regain, and describe changes in subjective appetite following a mixed-meal tolerance test (Exploratory).

DETAILED DESCRIPTION:
The TWIST 2.0 Study is a 12-month, 2-arm RCT in adults with recent weight loss. We will examine the efficacy of TRE on weight (Aim 1a) and fat mass (Aim 1b) regain, and describe changes in subjective appetite following a mixed-meal tolerance test (Exploratory). Potential participants will be screened via telephone and eligible participants will attend an in-person screening visit where they will complete questionnaires and have their height and weight measured. We will perform a 4-week run-in period to establish weight stabilization and measure eating patterns before randomization. Eligible participants following the run-in period will be randomized with equal allocation to one of the 2 arms: 1) TRE intervention ≤10-hr/day TRE intervention); or 2) CON. At baseline, 6 and 12 month measurements, participants will complete a bioelectrical impedance analysis (BIA) and dual energy x-ray absorptiometry (DEXA) scan by a certified radiology technician. Within each arm, participants will be randomized to either complete or not complete a mixed meal tolerance test in which they will consume a small portion of a protein shake and complete a visual analog scale (VAS) on their subjective hunger/fullness. Participants in both arms will receive one-page handouts (i.e., "advice") on topics to assist with weight maintenance. The only between-group differences are the TRE arm will be instructed to follow a restricted eating window of ≤10 hr/day, self-monitor foods and beverages into a smartphone app, measure body weight using a Bluetooth-enabled scale, and receive behavioral counseling directed at sustaining adherence to the TRE intervention. The CON arm will be unrestricted in their eating window and encouraged to eat a habitual breakfast, lunch, and dinner. No additional contact will be made between the CON arm and interventionist during the 12 months unless we schedule a measurement visit. Digital newsletters will be provided every month for the first 6 mos, and then every other month containing complementary information on WLM to engage participants in the CON arm. The same newsletters will be going to the TRE.

ELIGIBILITY:
Inclusion Criteria:

* ≥5% non-surgical weight loss in the last 3 mos;
* current BMI 20.5-45 mg/kg2;
* between the ages 25 to 65 years old;
* own a smartphone or willing to use a smartphone if provided for self-monitoring. For in-person screening, eligible participants will provide signed informed consent and have their temporal eating patterns measured.

Exclusion Criteria:

* pregnant, trying to get pregnant or breastfeeding;
* previous or planned bariatric surgery;
* previous or current history of eating disorder;
* ongoing participation in another weight-management research study;
* continued participation in a weight loss program other than the proposed study;
* currently on appetite suppressants;
* currently following intermittent fasting; or skipping meals;
* eating window <11h 59min/day;
* perform overnight shift work more than once a week;
* work that includes travel across one or more time zones;
* taking medications that affect body weight or would preclude TRE;
* unable or unwilling to provide informed consent;
* unable to participate meaningfully in the intervention (e.g., uncorrected sight and hearing impairment);
* unwilling to accept randomization assignment;
* unable to log at least 2 meals into the smartphone app for 70% (~20 days) during of the run-in period;
* have type 1 or type 2 diabetes, or other conditions that would preclude restricted eating windows;
* narcolepsy,
* >2.5 kg additional weight loss during run-in phase (weight regain is not an exclusion criteria);
* is non-English speaking (the mCC app is currently only available in English).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Absolute Body Weight Change | Baseline, Month 6, Month 12
Percent Body Weight Change | Baseline, Month 6, Month 12
Percentage of Participants with Successful Weight Loss-Maintenance (WLM) | Baseline, Month 6, Month 12
  WLM defined as regaining ≤25% of initial weight loss.
Absolute Fat Mass Change Measured with DEXA | Baseline, Month 6, Month 12
  Assessed using dual-energy x-ray absorptiometry (DEXA) scan.
Percent Fat Mass Change Measured with DEXA | Baseline, Month 6, Month 12
  Assessed using dual-energy x-ray absorptiometry (DEXA) scan.

OTHER OUTCOMES:
Incremental Area Under the Curve (iAUC) for appetite using a Visual Analog Scale (VAS) | Baseline, Month 6, Month 12
  The VAS allows participants to rate their appetite on a Likert scale from 1-10.

CONTACTS AND LOCATIONS:
Overall Officials: Collin Popp, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: collin.popp@nyulangone.org and margaret.curran@nyulangone.org. The protocol, statistical analysis plan and ICF will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposes to use the data will be granted access upon reasonable request. Requests should be directed to collin.popp@nyulangone.org and margaret.curran@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.